CLINICAL TRIAL: NCT03366246
Title: A Double-blind, Monocentric, Phase 3 Clinical Study for the Evaluation of Efficacy of a Topical Anesthetic Containing Lidocaine 25mg/g and Prilocaine 25mg/g in Adult Patients of Phototypes I to III in Treatment With CO2 Fractional Laser
Brief Title: Efficacy of a Topical Anesthetic Containing Lidocaine and Prilocaine in Treatment With CO2 Fractional Laser
Acronym: CO2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galeno Desenvolvimento de Pesquisas Clínicas (Other Government)
Collaborators: Biolab Sanus Farmaceutica (Industry)
Responsible Party: Principal Investigator, Gilberto De Nucci, PhD, Director and Principal Investigator, Galeno Desenvolvimento de Pesquisas Clínicas
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GDN 051/13
Record Dates: First submitted 2017-11-22; First posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Lidocaine Adverse Reaction; Prilocaine Adverse Reaction
Keywords: topical anesthetic; nanocapsules; nanotechnology; lidocaine; prilocaine; fractional CO2 laser resurfacing
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: Double-blind, crossover study where the same participant received in one side of the forehead the active drug and in the other side of the forehead placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: 1 tube containing anesthetic and 1 tube containing placebo, both with the same aspect (same vehicle) were randomized in respect of which side each formulation should be applied. Tubes were labeled with the subject number and the indication of LEFT or RIGHT side for application. Therefore, these identical tubes, no longer possible to distinguish whether a particular tube was referring to test or control formulation. Those responsible for the separation did not participate in the conduct of activities of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lidocaine / prilocaine cream (Active Comparator): according to randomization 2g topical nano anesthetic ( lidocaine 25mg/g and prilociane 25mg/g )was applied to one side ( left or right ) of the forehead 20 minutes before laser therapy.
  Interventions: Drug: Lidocaine / Prilocaine Cream
- placebo (Placebo Comparator): according to randomization 2g of the placebo( nano anesthetic vehicle with no active ingredient ) was applied to one side ( left or right) of the forehead 20 minutes before laser therapy.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Lidocaine / Prilocaine Cream — according randomized this side received placebo or active product
  Arms: lidocaine / prilocaine cream
Drug: placebo — according randomized this side received placebo or active product
  Arms: placebo

SUMMARY:
This is a study aimed at evaluating the efficacy of a topical anesthesia (test product) compared to placebo in adult patients of phototypes I to III, with indication of treatment of CO2 fractional laser in the forehead. In addition to efficacy, safety and tolerability of the product have been studied.

The product under investigation is a topical formulation containing lidocaine 25 mg/g and prilocaine 25mg/g which in previous studies performed in the same institution with healthy subjects in adulthood showed faster onset than other formulations. In these previous studies, the product was well tolerated, and there were no signs of a skin reaction or adverse events of a systemic nature.

The CO2 fractional laser treatment is routinely used by plastic surgery and dermatology for treatment with aesthetic purposes of skin imperfections. It's a procedure until certain painful point, which as a rule is performed without prior use of topical anesthetic.

The test product is believed to produce a clinically significant reduction of pain when compared to placebo, during the application of CO2 laser on the forehead for the aesthetic treatment of the face.

DETAILED DESCRIPTION:
The study was designed to allow assessing the efficacy of the product compared to placebo when applied to reduce pain resulting from treatment of the forehead with CO2 fractional laser at 5 mJ fluency and 5% concentration. To assess possible reactions, the photographic records were taken prior to the application of both products, as well as immediately prior to laser therapy and after 1 hour of laser therapy (1:20 h of application of the products).

In addition to the efficacy evaluation, the concomitant application of the control product (placebo) aimed to verify if possible dermatological reactions would be related to the active principle of the product or to the components of the cream base or to the performance of the laser therapy. In addition, considering a subgroup of participants, the study allowed the assessment of the degree of systemic absorption from the plasma concentrations observed, through the collection of blood samples for quantification of the compounds after their topical application.

Phase III, double-blind, monocentric, randomized crossover at the same time (right and left sides of forehead) , consisting of 120 patients, phototypes I to III, older than 18 years, female or male, with indication of aesthetic treatment with carbon dioxide (CO2) fractional laser in the forehead.

The anesthetic formulation, the object of the study, was administered topically in one side of the forehead and the placebo formulation (vehicle of the product) in the opposite side, once, as randomized, twenty minutes before the start of the CO2 laser therapy (in both sides of the forehead).

A total of 120 samples (5 g tubes) of the Test formulation and 120 samples (5 g tubes) of the Control (placebo) formulation were prepared for the administration of the medication to study . Initially, based on identification only on the secondary packaging (labeled plastic bag containing only test formulation tubes and labeled plastic bag containing only control formulation tubes), the tubes of each formulation were labeled with the subject's subject number and the indication of the side ( left or right ) of application, according to randomization of the study. After labeling and proper conferencing, these identical looking tubes were assembled and sorted by the participant number and left or right , and it was no longer possible to distinguish whether a particular tube concerned the test or control formulation. This set of samples was forwarded for conducting the study. Those responsible for the separation did not participate in the conduct of the study activities.

The study population consisted of female or male patients, phototypes I to III, with good general health conditions and those older than 18 years who had indication of aesthetic treatment with CO2 fractional laser compatible with the study proposal . These patients attended the clinic either spontaneously.

The anesthetic formulation and placebo were weighed individually, 2g of each gel, placing them directly on a spatula identified as left or right side, on a semi-analytical scale. The contents on the spatulas were applied to the corresponding forehead side using the gloved finger of the applicator to spread it as evenly as possible, 20 minutes before the session with CO2 fractional laser, under the supervision of the clinical investigator. Both test product and placebo gel were removed with saline solution and then CO2 laser intensity of 5mJ and concentration of 5% was applied across the forehead, always starting the right side toward the left side.

Immediately (0 min) after laser application and at 30, 60 and 90 minutes, it was assessed pain sensation in four quadrants of each forehead side using a visual analogue scale. The scale consists of a continuous line, whose left end corresponding to the absence of pain ("No Pain") and right end corresponding to the worst pain bearable by the patient ("the worst pain you can imagine"). The patient scored a perpendicular mark anywhere on the line (including the ends) in position to understand better represent the intensity of pain experienced on that quadrant at the specific time of each evaluation.

The evaluations were completed after 90 minutes of laser session (110 minutes after treatment with the investigational products) and blood pressure, pulse and temperature measurements were performed before the patient was released. At the end of the study, the distance from the left end to the mark was measured with a millimeter scale ruler. Two independent persons performed this measurement and any discrepancies values were conferred by a third person.

At the end of the procedure was generated a table in Excel, also conferred with the values obtained in centimeters for each occasion, including the total length of the ruler. The value in percentage was obtained by dividing the measured value by the total length of the scale by 100 . The averaged response corresponding to the four quadrants on the left and the average of the responses corresponding to the four quadrants on the right was calculated.

The two values (mean of the left side and mean of the right side) obtained for each of the occasions was the value used for the statistical calculation of treatment efficacy. A mean reduction of 30% with the topical anesthetic versus placebo - test / placebo ≤0.7 was considered clinically significant . The statistical analysis used for efficacy was the paired t-test.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male patients with phototypes I to III and older than 18 years and less than 70 years;
2. Indication of aesthetic treatment with CO2 fractional laser in the forehead;
3. Absence of treatment in the forehead that, at the discretion of the clinical investigator, may interfere with the objectives of the study;
4. Absence of allergic skin reactions on the face;
5. Lack of other significant diseases that, according to the criteria defined in this protocol, may be impacted by the medical criteria, and the evaluations to which it was submitted: clinical history, physical examination, ECG;
6. Capable of understanding the nature and purpose of the study, including risks and adverse effects, and intending to cooperate with the researcher and to act according to the requirements of the entire study, by signing the Informed Consent Form.

Exclusion Criteria:

1. The volunteer has known hypersensitivity to chemically related compounds; history of serious adverse reactions or hypersensitivity to any drug;
2. Known hypersensitivity to lidocaine, prilocaine, vehicle of the investigational product (gel) or to chemically related compounds; history of serious adverse reactions;
3. History of congenital or idiopathic methemoglobinemia
4. Current evidence of clinically significant diseases of gastrointestinal, cardiovascular, hepatic, renal, pulmonary, or other origin that prevent patient participation in the study and / or, at the discretion of the clinical investigator, expose the patient to additional risk ;
5. History of alcohol or drug abuse;
6. Treatment, within 3 months prior to the study, with any drug known to have a well-defined toxic potential in large organs;
7. Participation in any experimental study or ingestion of any experimental drug within six months prior to the start of this study; 8 .Positive pregnancy test , delivery or abortion in the 12 weeks prior to the scheduled start of treatment; 9 .Any condition that prevents the patient from participating in the study, according to the researcher's criteria.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-06-07 (Actual); Primary Completion 2014-07-25 (Actual); Study Completion 2014-07-25 (Actual)

PRIMARY OUTCOMES:
Pain assessed by means of a visual analog scale | at 0 minutes after laser therapy with CO2 fractional laser.
  The aim of this present study was to evaluate the efficacy of this new product compared to placebo when applied to the forehead of patients submitted to fractional CO2 laser, using a visual analog scale (VAS).The scale consists of a continuous line, whose left end corresponding to the absence of pain ("No Pain") and right end corresponding to the worst pain bearable by the patient ("the worst pain you can imagine"). The patient scored a perpendicular mark anywhere on the line (including the ends) in position to understand better represent the intensity of pain experienced on that quadrant at the specific time of each evaluation
Pain assessed by means of a visual analog scale | at 30 minutes after laser therapy with CO2 fractional laser.
  The aim of this present study was to evaluate the efficacy of this new product compared to placebo when applied to the forehead of patients submitted to fractional CO2 laser, using a visual analog scale (VAS).The scale consists of a continuous line, whose left end corresponding to the absence of pain ("No Pain") and right end corresponding to the worst pain bearable by the patient ("the worst pain you can imagine"). The patient scored a perpendicular mark anywhere on the line (including the ends) in position to understand better represent the intensity of pain experienced on that quadrant at the specific time of each evaluation.
Pain assessed by means of a visual analog scale | at 60 minutes after laser therapy with CO2 fractional laser
  The aim of this present study was to evaluate the efficacy of this new product compared to placebo when applied to the forehead of patients submitted to fractional CO2 laser, using a visual analog scale (VAS).The scale consists of a continuous line, whose left end corresponding to the absence of pain ("No Pain") and right end corresponding to the worst pain bearable by the patient ("the worst pain you can imagine"). The patient scored a perpendicular mark anywhere on the line (including the ends) in position to understand better represent the intensity of pain experienced on that quadrant at the specific time of each evaluation.
Pain assessed by means of a visual analog scale | at 90 minutes after laser therapy with CO2 fractional laser
  The aim of this present study was to evaluate the efficacy of this new product compared to placebo when applied to the forehead of patients submitted to fractional CO2 laser, using a visual analog scale (VAS).The scale consists of a continuous line, whose left end corresponding to the absence of pain ("No Pain") and right end corresponding to the worst pain bearable by the patient ("the worst pain you can imagine"). The patient scored a perpendicular mark anywhere on the line (including the ends) in position to understand better represent the intensity of pain experienced on that quadrant at the specific time of each evaluation.

SECONDARY OUTCOMES:
Adverse Event Incidence | at 0:50, 1:20 and 1:50 minutes after cream application
  As secondary objective were to evaluate the safety of possible dermatological reactions

OTHER OUTCOMES:
Lidocaine and Prilocaine Plasma Concentration | 0 - 12 hours
  Eight of the 120 participants also took part in blood sampling for dosing plasma concentrations from blood samples taken at 0:00, 0:10, 0:20, 0:30, 0:40, 0:50, 1:00, 1:10, 1:20, 1:30, 1:40, 1:50, 2:00, 2:20, 2:40, 3:00, 3:30, 4:00, 5:00, 6:00, 7:00, 8:00, 10:00 and 12:00 hours after the application, in order to characterize the general pharmacokinetic profile

CONTACTS AND LOCATIONS:
Overall Officials: Gilberto De Nucci, MD, Study Director — Galeno Desenvolvimento de Pesquisas Clinicas Ltda. - ME
Locations (1):
- Clinica Gobbato de Medicina e Dermatologia, Rio Claro, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
study protocol results